CLINICAL TRIAL: NCT01680081
Title: Adenosine-induced Stress Dynamic Myocardial Perfusion Imaging With Dual-source CT
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Slow recruitment of target subjects and difficulty registering subjects
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 1-2011-0064
Record Dates: First submitted 2012-09-03; First posted 2012-09-06 (Estimated); Last update posted 2019-01-23 (Actual); Status verified 2019-01

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- CT perfusion group (Experimental)
  Interventions: Other: Adenosine stress dynamic CT perfusion

INTERVENTIONS:
Other: Adenosine stress dynamic CT perfusion

SUMMARY:
This study was designed as a prospective multicenter trial to determine the accuracy of combined CT coronary angiography and perfusion imaging, specifically quantitative dynamic perfusion imaging in patients with suspicious coronary artery disease compared conventional coronary angiography and quantitative dynamic perfusion MRI as standard reference.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women patients, with age ranging 40-80.
2. Suspected coronary artery disease who are supposed to undergo invasive coronary angiography with appropriate clinical indications
3. Patients who are willing to sign the informed consent form

Exclusion Criteria:

1. Contraindication of CT Known allergy to iodinated contrast media or history of contrast-induced nephropathy Decreased renal function: elevated serum creatinine(>1.5mg/dl) Contraindication to beta-blockers Severe arrhythmia: arterial fibrillation or uncontrolled tachyarrhythmia, or advanced atrioventricular block (second or third degree heart block)
2. Contraindication of MRI Claustrophobia Metallic hazards Pacemaker implant eGFR<30 ml/min
3. Unstable or uncooperative patients
4. Limited life expectancy due to cancer or end-stage renal or liver disease
5. Evidence of severe symptomatic heart failure (NYHA Class III or IV)
6. Previous myocardial infarction, coronary artery intervention, coronary artery bypass surgery, or other cardiac surgery

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2012-01-30 (Actual); Primary Completion 2016-07-11 (Actual); Study Completion 2016-07-11 (Actual)

PRIMARY OUTCOMES:
Diagnostic accuracy of stress induced CT perfusion | 10-30 days
  Diagnostic accuracy of combined stress and rest dynamic CT perfusion and coronary angiography with dual x-ray sources in detection of hemodynamically significant stenosis of coronary artery compared with conventional coronary angiography and perfusion MRI in patients with suspicious coronary artery disease.

CONTACTS AND LOCATIONS:
Locations (1):
- Severance hospital, Seoul, South Korea